CLINICAL TRIAL: NCT06459752
Title: Combined Effects of Visceral Manipulation and Noble Technique on Inter-rectal Distance, Low Back Pain and Functional Disability in Post-partum Females With Diastasis Recti.
Brief Title: Combined Effects of Visceral Manipulation and Noble Technique on Post-partum Females With Diastasis Recti
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0564
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Diastasis Recti
Keywords: Diastasis recti; Low back pain; Post partum females; Visceral manipulation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): This group received three sessions a week for six weeks, with 30 minutes per session given to visceral manipulation and noble technique (15 minutes each technique).
  Interventions: Other: visceral manipulation and noble technique
- Group B (Active Comparator): This group receives three sessions a week for six weeks, with 15 minutes per session in which noble technique is applied.
  Interventions: Other: noble technique

INTERVENTIONS:
Other: visceral manipulation and noble technique — First, the patient will lie face-up on a massage or exam table. Physiotherapists feel viscera, major internal organs located in the abdomen by lightly pressing through abdominal muscles. Physiotherapist manual poking, pressing, and massage actions do three things:
  1. Reveals visceral adhesions.
  2. Find tender spots.
  3. Breaks up adhesions. Massaging and pressing stretch the collagen fibers that makeup fascia, which loosens tightly bound fibers to break up adhesions. This releases the organs and allows them to move more freely.
  Minor adhesions may resolve after one session. Tough, stubborn adhesions may require several sessions plus self-manipulation between sessions
  Arms: Group A
Other: noble technique — The patient is positioned in supine with both knees bent and feet flat on a firm surface. The patient then places her crossed hands over her abdomen to support and pull the rectus abdominis muscles towards the midline. Finally, the patient is asked to slowly raise her head until a slight contraction is felt in the abdomen, holding for 20 seconds and repeating the exercise up to 20 times a day
  Arms: Group B

SUMMARY:
Diastasis recti is characterized by an abnormal expansion of the gap between the medial sides of the rectus abdominis muscle and a lengthening of the linea alba (increased inter-recti distance). It is mainly caused by excessive intra-abdominal pressure. The abdominal muscles and connective structures expand from the growing uterus during pregnancy. Low back pain is a prevalent complaint that can result from various factors, including weakened core muscles and functional disability. The aim of the study would assess of combined effect of visceral manipulation and noble technique on Inter-rectal distance, low back pain and functional disability in post-partum females with diastasis recti.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted in DHQ Hospital Toba Tek Singh. A nonprobability convenience sampling technique will be used. There will be 34 participants. Participants will meet with inclusion criteria and be divided into two groups A and B. In Group A 17 participants will receive visceral manipulation technique with noble technique for 30 minutes per session, three sessions per week for 6 weeks. While in Group B 17 participants will just receive noble technique exercises for 15 min per session, three sessions per week for 6 weeks. Participants will be assessed before and after treatment through; Digital nylon calipers for diastasis recti, NPRS for pain, and Quebec Back Pain Disability Scale (QBPDS) to assess LBP-related functional. Data will be analyzed during SPSS software version 21

ELIGIBILITY:
Inclusion Criteria:

* Age between 22 to 35.
* Primiparous women with vaginal delivery and an IRD of >2 cm.
* Three to six months postpartum with the presence of diastasis rectus abdominis.
* Patients having moderate low back pain in NPRS.

Exclusion Criteria:

* Acute Malignancy
* Recent Abdominal or Pelvic surgery
* Having undergone spinal surgery in the previous six months
* Serious spinal pathology
* Serious cardiovascular or metabolic disease Pregnancy
* Herniation pain

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity.
Enrollment: 30 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Pain: NPRS | 6th week
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). Cronbach's alpha value of NPRS is 0.88
disability: Quebec Back Pain Disability Scale (QBPDS) | 6th week
  The Quebec Back Pain Disability Scale (QBPDS) measures the extent to which people with low back pain have difficulty with everyday activities. The questionnaire is composed of 20 items on daily activities. The items were selected from 6 relevant subdomains of functional skills for patients with low back pain.
Muscle separation: Digital nylon calipers | 6th week
  The Digital nylon calipers are a valid tool for measuring IRD above the umbilicus. For the caliper measurements with the abdominal muscles at rest, the participant was positioned in hook-lying, arms down by the side, with 1 pillow placed beneath the head. The examiner palpated the medial borders of the right and left rectus abdominis muscle bellies at the marked locations. The inside measurement jaws of the digital nylon calipers were positioned at the locations of the palpating fingers. The intra-class correlation coefficient values exceeded 0.75 for the digital calipers.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Neelam, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital Toba Tek Singh, Toba Tek Singh, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akram J, Matzen SH. Rectus abdominis diastasis. J Plast Surg Hand Surg. 2014 Jun;48(3):163-9. doi: 10.3109/2000656X.2013.859145. Epub 2013 Nov 21. PMID 24256310
- [Background] Arslan OE. Anatomy of the abdominal wall. Aesthetic surgery of the abdominal wall: Springer; 2005. p. 1-28.
- [Background] Flament JB, Avisse C, Delattre JFJAwhp, management. Anatomy of the abdominal wall. 2001:39-63.
- [Background] Grevious MA, Cohen M, Shah SR, Rodriguez P. Structural and functional anatomy of the abdominal wall. Clin Plast Surg. 2006 Apr;33(2):169-79, v. doi: 10.1016/j.cps.2005.12.005. PMID 16638461
- [Background] Cavalli M, Aiolfi A, Bruni PG, Manfredini L, Lombardo F, Bonfanti MT, Bona D, Campanelli G. Prevalence and risk factors for diastasis recti abdominis: a review and proposal of a new anatomical variation. Hernia. 2021 Aug;25(4):883-890. doi: 10.1007/s10029-021-02468-8. Epub 2021 Aug 6. PMID 34363190
- [Background] Gilleard WL, Brown JM. Structure and function of the abdominal muscles in primigravid subjects during pregnancy and the immediate postbirth period. Phys Ther. 1996 Jul;76(7):750-62. doi: 10.1093/ptj/76.7.750. PMID 8677279
- [Background] Brahmandam G, Lipsett BJ. Anatomy, Abdomen and Pelvis: Umbilical Cord. 2025 Jul 26. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557389/ PMID 32491321
- [Background] Benjamin DR, van de Water AT, Peiris CL. Effects of exercise on diastasis of the rectus abdominis muscle in the antenatal and postnatal periods: a systematic review. Physiotherapy. 2014 Mar;100(1):1-8. doi: 10.1016/j.physio.2013.08.005. Epub 2013 Oct 5. PMID 24268942
- [Background] Doubkova L, Andel R, Palascakova-Springrova I, Kolar P, Kriz J, Kobesova A. Diastasis of rectus abdominis muscles in low back pain patients. J Back Musculoskelet Rehabil. 2018 Feb 6;31(1):107-112. doi: 10.3233/BMR-169687. PMID 28946525